CLINICAL TRIAL: NCT02343159
Title: A Multicenter, Open-label Phase IV Study to Evaluate Whether a Medication Event Monitoring System (MEMS®) Can Improve Adherence to Tecfidera® (Delayed-release Dimethyl Fumarate) Treatment in Multiple Sclerosis Patients.
Brief Title: Study to Evaluate Whether a Medication Event Monitoring System (MEMS) Can Improve Adherence to Tecfidera Treatment in Multiple Sclerosis Patients.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 109MS413
Record Dates: First submitted 2015-01-09; First posted 2015-01-21 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Standard MEMS Cap (Experimental): A standard MEMS cap that records the time and date when the bottle is opened without a visual LCD reader. Standard-of-care commercial supply of DMF (BID oral capsule) will be used in this study.
  Interventions: Drug: dimethyl fumarate; Device: Medication Event Monitoring System (MEMS)
- Arm 2: Smart MEMS Cap (Experimental): A smart MEMS cap with feedback (an LCD reader that allows the participant to monitor DMF bottle openings). Standard-of-care commercial supply of DMF (BID oral capsule) will be used in this study.
  Interventions: Drug: dimethyl fumarate; Device: Medication Event Monitoring System (MEMS)
- Arm 3: Smart MEMS Cap + Counseling (Experimental): A smart MEMS cap with feedback (an LCD reader that allows the participant to monitor DMF bottle openings) and an adherence counseling intervention. Standard-of-care commercial supply of DMF (BID oral capsule) will be used in this study.
  Interventions: Drug: dimethyl fumarate; Device: Medication Event Monitoring System (MEMS); Behavioral: Adherence counseling

INTERVENTIONS:
Drug: dimethyl fumarate — 120 mg and 240 mg delayed release capsules
  Other Names: Tecfidera; DMF; BG000012
Device: Medication Event Monitoring System (MEMS) — The MEMS automatically compiles drug dosing history data by electronically recording the date and time of each opening of the medication container
Behavioral: Adherence counseling — A telephone call to discuss adherence and individualized strategies based on data collected via smart device (i.e., LCD reader)
  Arms: Arm 3: Smart MEMS Cap + Counseling

SUMMARY:
The primary objective of the study is to determine whether a Medication Event Monitoring System (MEMS®) cap with a liquid crystal display (LCD) reader (a "smart" cap) along with additional patient counseling intervention (Arm 3) can improve adherence to dimethyl fumarate (DMF) treatment in Multiple Sclerosis (MS) patients as compared to a MEMS cap without an LCD reader (a "standard" cap) and no patient counseling intervention (standard of care, Arm 1) at Month 12.

The secondary objectives of this study in this study population are: to determine if data display on a smart MEMS cap with an LCD reader (Arm 2) can improve adherence as compared to a standard MEMS cap without an LCD reader (Arm 1) at Month 12; to determine whether the addition of patient counseling intervention based on MEMS data (Arm 3), or data display from a MEMS cap with an LCD reader (Arm 2) can improve adherence compared to standard MEMS cap without an LCD reader (Arm 1) at Month 6; to assess persistence and compliance at Months 6 and 12 for all arms; to assess the association between adherence and patient- reported outcomes (PROs) for all arms including Multiple Sclerosis Impact Scale (MSIS-29), and the Work Productivity and Activity Impairment Questionnaire (WPAI): MS v2.0.

ELIGIBILITY:
Key Inclusion Criteria:

* The candidate is a DMF-naïve patient
* Have a diagnosis of relapsing forms of MS and satisfy the approved therapeutic indication for DMF
* Have a recent (i.e., within the previous 6 months) complete blood count with results that do not preclude the patient's participation in the study, in the judgment of the Investigator

Key Exclusion Criteria:

* Have comorbid conditions that preclude participation in the study, as determined by the Investigator
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity
* Are participating, planning to participate, or have participated in the Tecfidera QuickStart Program

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (29):
- United States (29):
  - Research Site, Homewood, Alabama
  - Research Site, Pheonix, Arizona
  - Research Site, Carlsbad, California
  - Research Site, Los Angeles, California
  - Research Site, Panorama City, California
  - Research Site, Sacramento, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Merrillville, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Akron, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Hodges, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Round Rock, Texas
  - Research Site, Winchester, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Started | 27 | 27 | 30
Completed | 1 | 1 | 0
Not Completed | 26 | 26 | 30
Not completed — Early Study Termination | 16 | 19 | 23
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Adverse Event | 4 | 4 | 2
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Enrollment Error | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population will be used for analysis. ITT is defined as all participants who were randomized and received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling | Total
Number analyzed (Participants) | 26 | 26 | 27 | 79
Age, Customized [Number; unit: Participants]
  18 - 50 Years | 21 | 19 | 17 | 57
  > 50 Years | 5 | 7 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 23 | 68
  Male | 4 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Adherence Rates at Month 12: Arm 3 vs. Arm 1
Description: Adherence is defined as the proportion of time on treatment over the study observation time period, times the proportion of actual DMF doses taken per label according to feedback from MEMS data over the total expected DMF doses per label during a treatment period.
Time Frame: Month 12
Population: The limited number of participants enrolled and the early termination of the study resulted in efficacy data not collected, and efficacy outcomes not analyzed, as per the pre-specified plan of analysis.
Arm/Group | Arm 1: Standard MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Adherence Rates at Month 12: Arm 2 vs. Arm 1
Description: as for outcome 1
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Adherence Rates at Month 6: Arm 3 vs. Arm 1
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Adherence Rates at Month 6: Arm 2 vs. Arm 1
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Persistence Rates at Months 6 and 12
Description: Persistence rates defined as the proportion of time on treatment over the study observation time period.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Compliance Rates at Month 6 and 12
Description: Compliance rates defined as the proportion of actual DMF doses taken per label according to feedback from MEMS data over total expected DMF doses per label during treatment period.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29)
Description: The 29-item MSIS-29 is a participant-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a participants perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI: MS Version 2.0)
Description: The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Month 6, Month 12
Population: as for outcome 1
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Collected between the time of informed consent and month 12 or early discontinuation visit.
Description: Safety population: Defined as all subjects who received at least one dose of study treatment.
Arm/Group | Arm 1: Standard MEMS Cap | Arm 2: Smart MEMS Cap | Arm 3: Smart MEMS Cap + Counseling
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/26 | 0/27
Other Adverse Events (participants affected / at risk) | 17/26 | 22/26 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Standard MEMS Cap (N=26) | Arm 2: Smart MEMS Cap (N=26) | Arm 3: Smart MEMS Cap + Counseling (N=27)
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Standard MEMS Cap (N=26) | Arm 2: Smart MEMS Cap (N=26) | Arm 3: Smart MEMS Cap + Counseling (N=27)
Fungal infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 2 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 9 | 10 | 8
Hot flush (Vascular disorders) | 0 | 1 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Transaminase increased (Investigations) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 4
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritis generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.